CLINICAL TRIAL: NCT04894253
Title: Study of the Immune Response to SARS-CoV-2 Vaccination in Patients With Systemic Lupus
Brief Title: Immune Response to SARS-CoV-2 Vaccination in Systemic Lupus
Acronym: LUPCELLVAX
Status: Terminated | Type: Observational
Why Stopped: inclusion difficulties
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 8263
Record Dates: First submitted 2021-05-18; First posted 2021-05-20 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Systemic Lupus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 18 Months
Biospecimen Retention: Samples Without DNA — Whole blood with subsequent extraction of:
  * Serum
  * Peripheral blood mononuclear cell
  * RNA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Single group of 30 patients with systemic lupus
  Interventions: Biological: SRAS-CoV-2 vaccination immunological response

INTERVENTIONS:
Biological: SRAS-CoV-2 vaccination immunological response — Follow for 18 months a single group of 30 patients with systemic lupus after their SRAS-CoV-2 vaccination.
  Intervention includes immunological analysis on additional volume of blood collected as part of routine care.

SUMMARY:
The main objective is to study the impact of vaccination against Covid-19 on the specific humoral and cellular immune response (against SARS-CoV-2) and non-specific (evolution of the pathological immune system of the disease), in a lupus population.

The secondary objective is to study the impact of lupus disease activity on the humoral and cellular response of patients following vaccination against SARS-CoV-2.

The hypothesis is that disease activity and / or certain treatments used in lupus may interfere with the humoral and cellular immune response induced by vaccination against SARS-CoV-2.

ELIGIBILITY:
Inclusion Criteria:

* Adult subject (≥ 18 years old), male or female
* Patient with systemic lupus according to ACR 1997 criteria
* Patient followed by the National Reference Center "Rare Systemic Autoimmune Diseases" of the University Hospitals of Strasbourg
* Patient who agreed to be vaccinated against SARS-CoV-2
* Subject having expressed his non-opposition to the research
* Subject affiliated to a social health insurance protection scheme

Exclusion Criteria:

* Patient treated by:

  * Corticosteroids (> = 10mg / day)
  * Immunosuppressant (azathioprine, mycophenolate mofetil, cyclophosphamide) to control lupus activity
  * A biomedicine targeting B cells (rituximab, belumimab).
* Inability to provide informed information about the subject (subject in an emergency, difficulty in understanding the subject, etc.)
* Subject under safeguard of justice
* Subject under guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with systemic lupus, monitored and vaccinated at the national reference center for "rare systemic autoimmune diseases" of the University Hospitals of Strasbourg.
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2021-06-07 (Actual); Primary Completion 2021-06-07 (Actual); Study Completion 2023-12-22 (Actual)

PRIMARY OUTCOMES:
Investigation of the immune response following vaccination against SARS-CoV-2 | 3 or 4 weeks
  Collection of clinical data and correlation with immunological analyzes of the biological samples
Investigation of the immune response following vaccination against SARS-CoV-2 | 3 months
  Collection of clinical data and correlation with immunological analyzes of the biological samples
Investigation of the immune response following vaccination against SARS-CoV-2 | 6 months
  Collection of clinical data and correlation with immunological analyzes of the biological samples
Investigation of the immune response following vaccination against SARS-CoV-2 | 12 months
  Collection of clinical data and correlation with immunological analyzes of the biological samples
Investigation of the immune response following vaccination against SARS-CoV-2 | 18 months
  Collection of clinical data and correlation with immunological analyzes of the biological samples

SECONDARY OUTCOMES:
Study the impact of lupus disease activity on SARS-CoV-2 vaccine immune response | 3 or 4 weeks
  Measurement of lupus disease activity by a validated score (SLEDAI) at the time of vaccination and follow-up.
Study the impact of lupus disease activity on SARS-CoV-2 vaccine immune response | 3 months
  Measurement of lupus disease activity by a validated score (SLEDAI) at the time of vaccination and follow-up.
Study the impact of lupus disease activity on SARS-CoV-2 vaccine immune response | 6 months
  Measurement of lupus disease activity by a validated score (SLEDAI) at the time of vaccination and follow-up.
Study the impact of lupus disease activity on SARS-CoV-2 vaccine immune response | 12 months
  Measurement of lupus disease activity by a validated score (SLEDAI) at the time of vaccination and follow-up.
Study the impact of lupus disease activity on SARS-CoV-2 vaccine immune response | 18 months
  Measurement of lupus disease activity by a validated score (SLEDAI) at the time of vaccination and follow-up.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital of Hautepierre, Strasbourg, Bas-Rhin, France